CLINICAL TRIAL: NCT00299689
Title: Phase II Trial of ONTAK With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James Graham Brown Cancer Center (Other)
Collaborators: University of Louisville (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 076.06
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2013-05

CONDITIONS: Malignant Melanoma
Keywords: Melanoma; Metastatic; Stage IV; Ontak
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — denileukin diftitox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention (Experimental): Single-arm: Ontak
  Interventions: Drug: Denileukin diftitox

INTERVENTIONS:
Drug: Denileukin diftitox — 12 mcg/kg IV (in vein) over 30 minutes on days 1 through 4 of each 21 day cycle for 4 cycles.
  Other Names: ONTAK

SUMMARY:
The purpose of this study is to determine whether ONTAK is an effective treatment in patients with Stage IV Melanoma

DETAILED DESCRIPTION:
This is a Phase II clinical trial to determine whether administration of ONTAK will result in a significant response rate in patients with metastatic melanoma.

Although the development of effective immunotherapy and the characterization of multiagent chemotherapy regimens have substantially improved in the treatment of metastatic malignant melanoma, the overall results remain dismal with a 6% five year survival rate for stage IV disease. Of the common adult-onset cancers, melanoma is widely held to be the most amenable to immunological intervention.

The primary objective of this study is to determine the response rate and the overall survival of patients with metastatic malignant melanoma treated with two regimens of ONTAK.

ELIGIBILITY:
Only patients with distant metastases from cutaneous or mucosal melanoma or melanoma of unknown primary are eligible for this study.

* Only patients with distant metastases from cutaneous or mucosal melanoma or melanoma of unknown primary are eligible for this study. All patients must fulfill the following criteria:

  * Primary tumor must be documented by histopathologic analysis
  * Measurable disease defined as at least one lesion that can be accurately and serially measured per the modified RECIST criteria (Appendix). Cutaneous lesions measuring at least 1 cm will be considered measurable. Measurements must be documented by radiologic examinations (CT scan, PET scan).
  * Disease recurrences occurring greater than five years after the original diagnosis must be biopsy proven.
  * Patients with lymph node metastases in multiple lymph node beds who are not amenable to surgical resection will be included in this study. Those patients with involvement of a single lymph node bed are not eligible.
* Liver Function: Patients must have adequate hepatic function documented by a serum bilirubin < 1.5 x the institutional upper limit of normal and liver enzymes (SGOT or SGPT and LDH and alkaline phosphatase) <2X the institutional upper limit of normal within 28 days prior to registration.
* Bone Marrow Function: Patients must have an absolute granulocyte count > 1,500/ul and platelet count > 100,000/ul obtained within 14 days prior to registration.
* Renal Function: Patients must have either a serum creatinine <1.5 mg/dl or a calculated creatinine clearance > 75 cc/min using the following formula:
* Estimated Creatinine Clearance = (140-age) X WT(kg) X 0.85 (if female 0.72) X creatinine (mg/dl) These tests must have been performed within 28 days prior to registration.
* Patients must have a MRI of the head performed within four weeks prior to registration.
* Cardiac Function: Patients must not have a history of ventricular fibrillation, sinus node or AV nodal disease, Wolff Parkinson White Syndrome, evidence of congestive heart failure, symptoms of coronary artery disease, serious cardiac arrhythmia, or evidence of prior myocardial infarction on EKG. The qualifying EKG must have been performed prior to study registration, but no earlier than 28 days prior to the definitive surgery. A normal cardiac stress test within 182 days prior to randomization is required for all patients over 50 years old or those with abnormal EKG or any history of cardiac disease.
* Patients must not have evidence of symptomatic pulmonary disease. PFT's within 182 days prior to registration showing a FEV1 > 2.0 liters or >75% of predicted are required for patients over 50 or with history of pulmonary symptoms.
* Patients with known autoimmune disorders, conditions of immunosuppression or treatment with systemic corticosteroids are not eligible for this study. Patients with known AIDS or HIV-1 associated complex or known to be HIV antibody seropositive are not eligible for this study.
* All patients must be 18 years of age or older.
* All patients must have a Zubrod Performance Status of 0 -1
* Patients must not be planning to receive concomitant other biologic therapy, radiation therapy, hormonal therapy, other chemotherapy, surgery, or other therapy while on this protocol.
* Pregnant or nursing women may not participate in this trial. Women/men of reproductive potential may not participate unless they have agreed to use an effective contraceptive method. A beta HCG pregnancy test is required within 14 days of registration for women of childbearing potential.
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-03; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chesney, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- James Graham Brown Cancer Center, Univ. of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Telang S, Rasku MA, Clem AL, Carter K, Klarer AC, Badger WR, Milam RA, Rai SN, Pan J, Gragg H, Clem BF, McMasters KM, Miller DM, Chesney J. Phase II trial of the regulatory T cell-depleting agent, denileukin diftitox, in patients with unresectable stage IV melanoma. BMC Cancer. 2011 Dec 13;11:515. doi: 10.1186/1471-2407-11-515. PMID 22165955
- [Derived] Rasku MA, Clem AL, Telang S, Taft B, Gettings K, Gragg H, Cramer D, Lear SC, McMasters KM, Miller DM, Chesney J. Transient T cell depletion causes regression of melanoma metastases. J Transl Med. 2008 Mar 11;6:12. doi: 10.1186/1479-5876-6-12. PMID 18334033

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Single-arm: Ontak
  Denileukin diftitox : 12 mcg/kg IV (in vein) over 30 minutes on days 1 through 4 of each 21 day cycle for 4 cycles.
Period: Overall Study
Arm/Group | Intervention
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 69
Age, Customized [Number; unit: Participants]
  >= 18 years | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Positive Response Defined as Clinical Complete Response, Partial Response or Stable Disease (Persisting for at Least 4 Weeks) as Measure by Modified RECIST Criteria
Time Frame: 2 weeks after completion of second cycle
Measure: Number; unit: participants
Arm/Group | Intervention
Number analyzed (Participants) | 16
participants | 16

2. Secondary Outcome: Overall Survival
Time Frame: All cause mortality
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes